CLINICAL TRIAL: NCT06011343
Title: Tofacitinib Associated With Meglumine Antimoniate in the Control of American Tegumentary Leishmaniasis. A Randomized and Controlled Clinical Trial.
Brief Title: Tofacitinib Associated With Meglumine Antimoniate in Cutaneous Leishmaniasis
Acronym: CLTofa23
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitário Professor Edgard Santos (Other)
Collaborators: Instituto Gonçalo Muniz FIOCRUZ BA (Unknown)
Responsible Party: Principal Investigator, Paulo Roberto Lima Machado, Senior Researcher, Hospital Universitário Professor Edgard Santos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL Tofa23
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Cutaneous Leishmaniasis, American
Keywords: Cutaneous Leishmaniasis, meglumine antimoniate, tofacitinib
MeSH Terms: conditions — Leishmaniasis, Mucocutaneous; Leishmaniasis, Cutaneous | interventions — tofacitinib

STUDY DESIGN:
Intervention Model Description: CL patients will be allocated in 2 intervention groups.
Who Masked: Participant, Investigator
Masking Description: After randomization and allocation each patient will receive a code that will be confidential.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo and Sbv (Placebo Comparator): Eleven CL patients will receive meglumine antimoniate by EV route at 20mg/kg/day, for 20 days.
  Interventions: Drug: Parenteral meglumine antimoniate
- Tofacitinib and Sbv (Experimental): Eleven CL patients will receive oral tofatinib (10mg daily for 30 days) associated to meglumine antimoniate by EV route at 20mg/kg/day, for 20 days.
  Interventions: Drug: Oral tofacitinib; Drug: Parenteral meglumine antimoniate

INTERVENTIONS:
Drug: Oral tofacitinib — Association of tofacitinib and meglumine antimoniate
  Arms: Tofacitinib and Sbv
Drug: Parenteral meglumine antimoniate — Meglumine antimoniate

SUMMARY:
Phase 2/3 randomized and controlled clinical trial, which will evaluate the effectiveness of the association meglumine antimoniate (Glucantime) with tofacitinib in the cure of CL and the capacity of this association to reduce the time of cure of the disease.

DETAILED DESCRIPTION:
1. STUDY AREA The southeastern region of the State of Bahia, Brazil, where the village of Corte de Pedra and adjacent towns are located, is one of the most important American Tegumentary Leishmaniasis (ATL) endemic area in Latin America. The Corte de Pedra Health Center, in the municipality of Tancredo Neves, is located 280km from Salvador and is a Reference Center for Diagnosis and Treatment of ATL. Yearly, more than 500 cases of patients with ATL are diagnosed and treated at this Center.

   The Health Center was established in 1986 and clinical physicians, dermatologists, otorhinolaryngologists and immunologists from the Immunology Service of the Federal University of Bahia, the Gonçalo Moniz Institute (IGM) and the Federal University of Recôncavo Bahiano (UFRB) visit the area every two weeks. The Post also has the support of 4 trained health agents, all residents of the region. They assist patients, visit families, and participate in research activities.
2. STUDY DESIGN

   A. Type of study:

   This project is a phase 2/3 randomized and controlled clinical trial, which will evaluate the effectiveness of the association meglumine antimoniate (Glucantime) with tofacitinib in the cure of CL. the main objectives are: 1. To compare the cure rate of meglumine antimoniate associated with tofacitinib with meglumine antimoniate alone in the treatment of CL caused by L. braziliensis; 2. To determine whether combined treatment with meglumine antimoniate associated with tofacitinib reduces CL healing time.

   B. Definition of cases:

   Cutaneous Leishmaniasis: Presence of a typical ulcerated lesion on the skin, without evidence of mucosal involvement, with a positive skin test and disease duration between 30 and 90 days. The diagnosis will be made by identifying amastigotes in the histopathological study with immunohistochemistry and/or documentation of DNA for L.braziliensis by polymerase chain reaction (PCR).

   C. Methodology:

   The rate of cure or treatment failure is only defined on day 90 after starting therapy. We estimate that combining Glucantime with tofacitinib will increase the healing rate and reduce the healing time of CL. The present proposal is a proof of concept with the participation of patients with CL with disease duration between 30 and 90 days and with ulcer size between 10 and 60mm. Patients will be randomized, group 1 will receive Glucantime at a dose of 20mg/Kg/weight /day with a maximum dose of 1200mg intravenously for 20 days, and group 2 will be treated with Glucantime at the dose and time period described above associated with tofacitinib at a dose of 10mg/day for 30 days. Patients will be evaluated on day 0, day 30, day 60 and day 90 to determine the size and characteristics of the ulcers and the occurrence of wound healing.

   Sample size calculation: Considering that healing of ulcers up to 60mm in diameter in patients with CL with Glucantime will occur in 50% of patients while the cure rate in patients receiving Glucantime combined with tofacitinib will be 90% with a power of 80% and P< 0.05, 22 patients will be needed, 11 in each group.

   Subjects will be allocated in the 2 study arms after randomization at www.randomization.com.
3. ETHICAL CONSIDERATIONS Participation in the study is voluntary and all participants must, after reading and understanding the nature of the study, benefits and risks, sign the attached Free and Informed Consent Form (TCLE). This study was approved by the ethics committee of the Faculty of Medicine of Bahia, Federal University of Bahia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with CL of both sexes with disease duration between 30 and 90 days. Patients with CL will be treatment-naïve for leishmaniasis. Individuals will be explained about the nature of the study and will only be included if they agree to participate and sign the Free and Informed Consent Form.

Exclusion Criteria:

* Patients under the age of 18 and pregnant women will not participate in the study considering the need to withdraw 30 ml of blood to carry out the studies of the immune response. Patients over 60 years old, debilitating chronic diseases such as heart failure, liver failure, kidney failure, HIV infection and use of immunosuppressant drugs will also not participate in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Cure at 90 days | 90 days
  Healing will be defined by complete healing of the ulcer and re-epithelialization of the skin on day 90, in the absence of infiltrated borders. Failure will be defined as persistence of the ulcer at day 90 with ulcer healing occurring but persistent infiltration at the edges.

SECONDARY OUTCOMES:
Cure at 180 days | 180 days
  Absence of relapse after 180 days
Time to cure | Days
  Time (in days) until complete healing of the ulcer and re-epithelialization of the skin in the absence of infiltrated borders.
Adverse events | 45 dyas
  Adverse events will be recorded and graded

CONTACTS AND LOCATIONS:
Overall Officials: EDGAR CARVALHO, MD, PhD, Principal Investigator — Federal University of Bahia
Locations (1):
- Corte de Pedra Health Post, Presidente Tancredo Neves, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.